CLINICAL TRIAL: NCT07137988
Title: Effect of Acute Grape Seed Extract Supplementation on the Heart Rate Recovery in Young Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Principal Investigator, Jong-Kyung Kim, Professor, California Baptist University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 034-2425-EXP
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Young Men
Keywords: Double blinded cross-over design
MeSH Terms: interventions — Grape Seed Extract; Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Heart rate recovery with grape seed extract (Experimental): Grape seed extract: 300 mg, two capsules Starch: 300 mg, two capsules
  Interventions: Dietary Supplement: 600 mg grape seed extract; Dietary Supplement: 600 mg Starch
- Sham Comparator: Experimental: BFR exercise without histamine blockade (Placebo Comparator): Heart rate recovery with placebo (starch, 300 mg, 2 capsules)
  Interventions: Dietary Supplement: 600 mg grape seed extract; Dietary Supplement: 600 mg Starch

INTERVENTIONS:
Dietary Supplement: 600 mg grape seed extract — Each participant took either GSE (300 mg, 2 capsules) or a placebo (300 mg, 2 capsules filled with starch) 2 hours before their scheduled lab visit. The supplements were made to look identical to prevent any bias from the participants or the testers. There was a washout period of at least 72 hours, but no more than a week, between each trial.
  Other Names: 600 mg starch
Dietary Supplement: 600 mg Starch — Each participant took either GSE (300 mg, 2 capsules) or a placebo (300 mg, 2 capsules filled with starch) 2 hours before their scheduled lab visit. The supplements were made to look identical to prevent any bias from the participants or the testers. There was a washout period of at least 72 hours, but no more than a week, between each trial.

SUMMARY:
This study hypothesized that sustained sympathoexcitation via MMA slows down PHRR and that GSE supplementation is effective at improving PHRR in young individuals. 12 Participants were randomly assigned, via a double-blind, cross-over design, to either receive GSE (300mg, 2 capsules) or PL (300mg, 2 capsules), with a washout period of at least 72 hrs. between trials. A submaximal exercise test was performed using a cycle ergometer combined with isometric handgrip exercise using a handgrip dynamometer, and blood flow occlusion by placing a cuff over the brachial artery of the dominant arm. Post heart rate recovery (PHRR) was measured at 5 sec. intervals throughout the experiment. The PHRR was evaluated between GSE and PL at every min. for 300 sec.

ELIGIBILITY:
Inclusion Criteria:

* good health, nonsmokers, those not taking medications that could affect cardiovascular function

Exclusion Criteria:

* hypertension, muscular skeletal disorders

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate recovery every minute and heart rate kinetics (tau) following exercise | 5 min after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided